CLINICAL TRIAL: NCT01498887
Title: A Multi-centre, Open-label, Non-randomised, Parallel Group Clinical Trial to Assess the Efficacy of Fingolimod in Naive Patients Versus Fingolimod in Patients Previously Treated With Interferons or Glatiramer Acetate, Based on the Presence of Relapses in Patients With Relapsing-remitting Multiple Sclerosis.
Brief Title: Efficacy of Fingolimod in de Novo Patients Versus Fingolimod in Patients Previously Treated With a First Line Disease Modifying Therapy
Acronym: EARLiMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DES03; 2011-003484-30 (EudraCT Number)
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Fingolimod; Early multiple sclerosis; Naive patients
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naive or de novo participants (Experimental): Participants received 0.5 mg FTY720 (fingolimod) orally once daily for 12 months.
  Interventions: Drug: Fingolimod (FTY720)
- Previously treated with first-line DMTs participants (Experimental): Participants received 0.5 mg FTY720 (fingolimod) orally once daily for 12 months.
  Interventions: Drug: Fingolimod (FTY720)

INTERVENTIONS:
Drug: Fingolimod (FTY720) — Hard gelatin capsules containing 0.5 mg of fingolimod.

SUMMARY:
This study assessed the efficacy of fingolimod in patients with short duration relapsing-remitting multiple sclerosis who had not been previously treated with disease-modifying therapies (DMTs), versus patients with the same disease duration who had previously received first-line DMTs.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple sclerosis, according to the 2010 revised McDonald criteria, with a relapsing-remitting course, and with at least 9 T2 lesions consistent with the disease, with disease duration greater than or equal to one year and less than or equal to five years.
* Patients who have had at least two relapses in the past two years and an Expanded Disability Status Scale score between 0 and 3.5, inclusive.

Patients

* Treatment naïve: patients who have never been treated with a Disease Modifying Therapy or
* Previously treated with a first-line Disease Modifying Therapy

Exclusion Criteria:

* Patients who have received treatment with:

Fingolimod at any time (e.g. participation in a fingolimod clinical trial), Immunosuppressant drugs such as azathioprine or methotrexate at any time; Immunoglobulins in the past 6 months. Monoclonal antibodies including natalizumab, Cladribine, cyclophosphamide or mitoxantrone, at any time.

- Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2011-12-24 (Actual); Primary Completion 2015-12-26 (Actual); Study Completion 2015-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- Australia (15):
  - Novartis Investigative Site, East Gosford, New South Wales
  - Novartis Investigative Site, Kanwal, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Bedford Park
  - Novartis Investigative Site, Brisbane Queensland
  - Novartis Investigative Site, Geelong VIC
- Spain (24):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, León, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, non-randomized, parallel group study.
Period: Overall Study
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Started | 200 | 147
Safety Set | 200 | 147
Intent-to-treat | 185 | 135
Completed | 184 | 136
Not Completed | 16 | 11
Not completed — Administrative problems | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Lack of Efficacy | 5 | 3
Not completed — Abnormal result from test procedure | 1 | 1
Not completed — Abnormal laboratory value | 2 | 2
Not completed — Adverse Event | 4 | 1

BASELINE CHARACTERISTICS:
Population: The analysis of the baseline characteristics was done on the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants | Total
Number analyzed (Participants) | 185 | 135 | 320
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.1 (8.08) | 34.0 (7.44) | 33.5 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 88 | 225
  Male | 48 | 47 | 95

OUTCOME MEASURES:

1. Primary Outcome: Annual Relapse Rate (ARR)
Description: ARR = 365 days * number of relapses / total days taking the study medication.
Time Frame: 12 months
Population: The ITT population was analyzed. The ITT consisted of all participants included in the safety population who met the inclusion/exclusion criteria and had at least one primary endpoint (ARR) measurement recorded.
Measure: Mean (Standard Deviation); unit: Relapses per year
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 185 | 135
Relapses per year | 0.290 (0.7399) | 0.354 (0.8547)
Statistical Analysis 1: Comparison: Naive or de Novo Participants vs Previously Treated With First-line DMTs Participants; Test type: Superiority or Other; p = 0.3118, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to First Relapse
Description: Time to first relapse was defined as the time from the first day of treatment to the first day of a new neurological symptom or worsening of an existing one.
Time Frame: first day of treatment to the first day of a new neurological symptom or worsening of an existing one, up to 12 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 185 | 135
months | NA [NA to NA] — Since less than half of the ITT population had a relapse, the median time since fingolimod treatment initiation to the first relapse was not reached. | NA [NA to NA] — Since less than half of the ITT population had a relapse, the median time since fingolimod treatment initiation to the first relapse was not reached.

3. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score
Description: The EDSS is an ordinal clinical rating scale ranging from a total score of 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. A negative change from baseline indicates improvement.
Time Frame: baseline, 12 months
Population: Participants from the ITT population with both baseline and 12 month values were analyzed. The ITT consisted of all participants included in the safety population who met the inclusion/exclusion criteria and had at least one primary endpoint (ARR) measurement recorded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 182 | 130
score on a scale | 0.000 (0.8040) | -0.077 (0.7911)

4. Secondary Outcome: Change From Baseline in Cerebral Volume
Description: Cerebral volume was assessed by magnetic resonance imaging (MRI). A negative change from baseline indicates improvement.
Time Frame: baseline, 12 months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 92 | 43
Percent change | -0.595 [-0.759 to -0.431] | -0.387 [-0.583 to -0.191]

5. Secondary Outcome: Percentage of Participants With Mild, Moderate or Severe Relapse
Description: The investigator classified a relapse as moderate-severe if oral or intravenous (IV) treatment (according to the local clinical practice) with steroids and/or hospitalization was needed. If neither oral nor IV treatment with steroids nor hospitalization was needed, the relapse was considered as mild.
Time Frame: 12 months
Population: Only participants from the ITT population with severity values were analyzed. The ITT consisted of all participants included in the safety population who met the inclusion/exclusion criteria and had at least one primary endpoint (ARR) measurement recorded.
Measure: Number; unit: Percentage of participants
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 47 | 39
Percentage of participants
  Mild | 42.55 | 38.46
  Moderate | 57.45 | 56.41
  Severe | 0.00 | 5.13

6. Secondary Outcome: Percentage of Relapse-free Participants
Description: Relapse-free participants were defined as participants who experienced no new neurological symptom or worsening of an existing one (relapses) during the 12-month treatment period with 0.5 mg fingolimod.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 185 | 135
Percent | 71.89 | 66.67

7. Secondary Outcome: Mean Number of T2 Active Lesions
Description: The mean number of new or enlarged T2 active lesions was assessed by MRI.
Time Frame: 12 months
Population: Participants from the ITT population with 12 month T2 lesion numbers were analyzed. The ITT consisted of all participants included in the safety population who met the inclusion/exclusion criteria and had at least one primary endpoint (ARR) measurement recorded.
Measure: Mean (Standard Deviation); unit: T2 lesions
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants
Number analyzed (Participants) | 163 | 106
T2 lesions | 2.0 (3.36) | 1.6 (2.72)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit, approximately 4 years.
Arm/Group | Naive or de Novo Participants | Previously Treated With First-line DMTs Participants | All Participants
Serious Adverse Events (participants affected / at risk) | 11/200 | 4/147 | 15/347
Other Adverse Events (participants affected / at risk) | 143/200 | 114/147 | 257/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naive or de Novo Participants (N=200) | Previously Treated With First-line DMTs Participants (N=147) | All Participants (N=347)
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 2
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 2 | 1 | 3
Partial seizures (Nervous system disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naive or de Novo Participants (N=200) | Previously Treated With First-line DMTs Participants (N=147) | All Participants (N=347)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 2
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 9 | 7 | 16
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Atrioventricular block first degree (Cardiac disorders) | 2 | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 1 | 2
Palpitations (Cardiac disorders) | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Retinal anomaly congenital (Congenital, familial and genetic disorders) | 1 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2
Amblyopia (Eye disorders) | 0 | 1 | 1
Astigmatism (Eye disorders) | 2 | 1 | 3
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 2
Diplopia (Eye disorders) | 2 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 1
Erythema of eyelid (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 1
Macular oedema (Eye disorders) | 1 | 0 | 1
Myopia (Eye disorders) | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Optic atrophy (Eye disorders) | 1 | 0 | 1
Pinguecula (Eye disorders) | 1 | 0 | 1
Presbyopia (Eye disorders) | 0 | 1 | 1
Retinal pigment epitheliopathy (Eye disorders) | 1 | 0 | 1
Strabismus (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 2 | 3 | 5
Visual impairment (Eye disorders) | 2 | 2 | 4
Vitreous floaters (Eye disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 8
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 1 | 1 | 2
Dental cyst (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 9 | 14
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2
Gastritis (Gastrointestinal disorders) | 3 | 1 | 4
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 4 | 1 | 5
Nausea (Gastrointestinal disorders) | 7 | 5 | 12
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 4 | 6
Adverse drug reaction (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 2
Chest pain (General disorders) | 1 | 3 | 4
Exercise tolerance decreased (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 11 | 9 | 20
Gait disturbance (General disorders) | 0 | 2 | 2
Influenza like illness (General disorders) | 1 | 1 | 2
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 5 | 6
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0 | 3
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 1 | 2
Ear infection (Infections and infestations) | 1 | 2 | 3
Folliculitis (Infections and infestations) | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 9 | 6 | 15
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Genital herpes (Infections and infestations) | 1 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 1
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 1 | 3
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 3 | 3 | 6
Laryngitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 3
Molluscum contagiosum (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 16 | 8 | 24
Onychomycosis (Infections and infestations) | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 1
Oral herpes (Infections and infestations) | 7 | 5 | 12
Paronychia (Infections and infestations) | 1 | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0 | 1
Pertussis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 8 | 4 | 12
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 4 | 2 | 6
Rhinitis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 5
Sinusitis bacterial (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 3 | 3
Tinea versicolour (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 6 | 3 | 9
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 2 | 2
Tooth infection (Infections and infestations) | 1 | 2 | 3
Tracheobronchitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 15 | 12 | 27
Urinary tract infection (Infections and infestations) | 15 | 15 | 30
Viral infection (Infections and infestations) | 3 | 0 | 3
Viral pharyngitis (Infections and infestations) | 1 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 2 | 5 | 7
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 2
Wound infection bacterial (Infections and infestations) | 1 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 4
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 3
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 5 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 5
B-lymphocyte count decreased (Investigations) | 1 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 1
Blood chloride increased (Investigations) | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 2 | 3
Blood iron decreased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 1 | 1 | 2
Blood triglycerides increased (Investigations) | 0 | 2 | 2
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 1
CD8 lymphocytes decreased (Investigations) | 1 | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 3
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 2 | 3
Micturition urgency (Investigations) | 0 | 1 | 1
T-lymphocyte count decreased (Investigations) | 1 | 0 | 1
Transaminases abnormal (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 1 | 2
Weight increased (Investigations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 4 | 16
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myokymia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1 | 1
Aphonia (Nervous system disorders) | 0 | 2 | 2
Balance disorder (Nervous system disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 7 | 12
Dysaesthesia (Nervous system disorders) | 1 | 1 | 2
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 17 | 17 | 34
Hemiparesis (Nervous system disorders) | 0 | 1 | 1
Hyperreflexia (Nervous system disorders) | 1 | 0 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 4
Lethargy (Nervous system disorders) | 1 | 0 | 1
Migraine (Nervous system disorders) | 6 | 6 | 12
Migraine with aura (Nervous system disorders) | 2 | 0 | 2
Migraine without aura (Nervous system disorders) | 2 | 0 | 2
Multiple sclerosis relapse (Nervous system disorders) | 2 | 1 | 3
Neuralgia (Nervous system disorders) | 2 | 0 | 2
Neurological symptom (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1
Optic neuritis (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 4 | 7
Partial seizures (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 2
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 2
Sensorimotor disorder (Nervous system disorders) | 1 | 0 | 1
Sleep paralysis (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 2 | 3
Syncope (Nervous system disorders) | 1 | 1 | 2
Tension headache (Nervous system disorders) | 1 | 1 | 2
Typical aura without headache (Nervous system disorders) | 1 | 0 | 1
Uhthoff's phenomenon (Nervous system disorders) | 1 | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 1
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 11 | 6 | 17
Anxiety disorder (Psychiatric disorders) | 1 | 1 | 2
Bruxism (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 1 | 2
Depression (Psychiatric disorders) | 9 | 6 | 15
Dysthymic disorder (Psychiatric disorders) | 1 | 1 | 2
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 5 | 3 | 8
Laziness (Psychiatric disorders) | 0 | 1 | 1
Personality disorder (Psychiatric disorders) | 2 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 2
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Acne (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Intraocular lens implant (Surgical and medical procedures) | 0 | 1 | 1
Skin lesion excision (Surgical and medical procedures) | 1 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.